CLINICAL TRIAL: NCT06427343
Title: The Effects of Low-dose Versus High-dose Intravenous Iron Therapy With Ferric Derisomaltose in Patients With Chronic Heart Failure and Iron Deficiency: a Randomized, Open-label, Blind Endpoint Trial (IRONDOSE)
Brief Title: The Effects of Low-Dose Versus High-Dose Intravenous IRON Therapy With Ferric DerisomaltOSE in Patients With Chronic Heart Failure and Iron Deficiency
Acronym: IRONDOSE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingyi Ren, Professor of medicine(Cardiology), Deputy Director of the Cardiology Department and Director of the Heart Failure Center, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-ZF-62
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Iron Deficiency
Keywords: IRONDOSE
MeSH Terms: conditions — Heart Failure; Iron Deficiencies | interventions — ferric derisomaltose

STUDY DESIGN:
Intervention Model Description: Drug: Ferric Derisomaltose
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose (Experimental): Participants randomized to this arm will receive repeat iron dosing as long as the serum ferritin was not >700 ng/mL, or if TSAT was not >40% during follow-up.
  Iron to be administered as ferric derisomaltose. Ferric derisomaltose will be administered according to the dosing schedule determined by the patient's body weight and hemoglobin value.
  Infused over a minimum of 15 mins for doses up to and including 1000mg, and a minimum of 30 mins for doses >1000mg.
  Interventions: Drug: High-dose ferric derisomaltose
- Low dose (Active Comparator): Participants randomized to this arm will receive repeat iron dosing if ferritin <100 ng/mL or if ferritin 100-300 ng/mL and TSAT <20% during follow-up.
  Iron to be administered as ferric derisomaltose in analogy to high-dose arm.
  Interventions: Drug: Low-dose ferric derisomaltose

INTERVENTIONS:
Drug: High-dose ferric derisomaltose — After baseline assessment, participants will be randomized in a 1:1 ratio to receive a high-dose IV iron regimen and a low-dose IV iron regimen. After the initial iron repletion, ferritin concentration and TSAT were measured every three months and the results used to determine the dose of ferric derisomaltose during follow-up.
  In the high-dose group, participants will receive repeat iron dosing as long as the serum ferritin was not >700 ng/mL, or if TSAT was not >40% during follow-up.
  Other Names: More intensive target
  Arms: High dose
Drug: Low-dose ferric derisomaltose — In the low-dose group, participants will receive repeat iron dosing if ferritin <100 ng/mL or if ferritin 100-300 ng/mL and TSAT >20% during follow-up.
  Other Names: Less intensive target
  Arms: Low dose

SUMMARY:
This study will address whether intravenous (IV) iron repletion with a more intensive target will provide greater benefits in improving exercise capacity for patients with chronic heart failure and iron deficiency. One group of participants will receive a high-dose IV iron regimen with a more intensive target, and the other group will receive a low-dose IV iron regimen with a less intensive target.

DETAILED DESCRIPTION:
Iron deficiency is a common and important comorbidity in heart failure. Randomized controlled trials have consistently demonstrated a beneficial effect of IV iron on exercise capacity and quality of life in iron-deficient patients with HF and reduced ejection fraction. However, these randomized controlled trials exhibit striking heterogeneity in targeting levels for maintenance strategies of IV iron repletion. Some studies (FERRIC-HF, FAIR-HF) withheld intravenous iron in cases of ferritin >800 ng/mL, hemoglobin >16.0 g/dL, or transferrin saturation (TSAT) >50%, while other studies (HEART-FID, IRONMAN) focused on targeting levels that are simply above the definition of iron deficiency. Additionally, the PIVOTAL trial showed that high-dose IV iron decreased recurrent heart failure events in patients undergoing hemodialysis compared to a lower-dose regimen. Whether functional outcomes differ between those on lower versus higher iron repletion targets among patients with heart failure remains unknown. This study will help us address this question.

This is an investigator-initiated, prospective, randomized, open-label blind endpoint study to assess the effects of high-dose IV iron repletion compared to a low-dose IV iron repletion on 12-month change in peak oxygen uptake (VO2) for patients with chronic heart failure and concomitant iron deficiency.

Patients with chronic heart failure and iron deficiency will be enrolled and randomized in a 1:1 ratio to receive a high-dose IV iron regimen and a low-dose IV iron regimen. After the initial iron repletion, ferritin concentration and TSAT were measured every three months and the results used to determine the dose of ferric derisomaltose during the follow-up period. In the high dose group, iron dosing will repeat as long as the serum ferritin was not >700ng/mL, or if TSAT was not >40%. Patients in the low dose group will receive repeat iron dosing if ferritin <100 ng/mL, or if ferritin 100-300 ng/mL and TSAT <20%, in line with criteria for iron deficiency in current guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Left ventricular ejection fraction (LVEF) <50% within 2 years prior to planned randomization (assessed by echocardiography or MRI).
3. New York Heart Association (NYHA) class II ~ III.
4. Either hospitalization for HF within 6 months prior to planned randomization or elevated plasma levels of natriuretic peptides within 3 months of randomization. a. For patients in sinus rhythm: NT- proBNP >300 pg/mL or BNP >100 pg/mL. b. For patients in atrial fibrillation: NT-proBNP >600 pg/mL or BNP >200 pg/mL.
5. Subjects with stable CHF (NYHA II/III functional class) on optimal background therapy (as determined by the investigator) for at least 4 weeks with no dose changes of heart failure drugs during the last 2 weeks (with the exception of diuretics).
6. Serum ferritin <100 ng/mL or serum ferritin 100-300 ng/mL and TSAT <20%.
7. Able and willing to perform a CPET at the time of randomization.
8. Able and willing to provide informed consent.

Exclusion Criteria:

1. Hemoglobin <9.0 g/dL or Hemoglobin >15.0 g/dL.
2. Renal dialysis or MDRD/CKD-EPI estimated glomerular filtration rate (eGFR) <15 ml/min/1.73m2.
3. Body weight <35 kg.
4. Heart failure was secondary to valvular diseases or congenital heart diseases.
5. History of acquired iron overload; known hemochromatosis or first relatives with hemochromatosis.
6. Known hypersensitivity to ferric derisomaltose or other IV iron product.
7. Known active infection (defined as currently treated with oral or intravenous antibiotics), bleeding (gastrointestinal hemorrhagia, menorrhagia, history of peptic ulcer with no evidence of healing or inflammatory bowel disease), malignancy, and hemolytic anemia.
8. History of chronic liver disease and/or alanine transaminase (ALT) or aspartate transaminase (AST) >3 times the upper limit of the normal range; myelodysplastic disorder; and known HIV/AIDS disease.
9. Acute myocardial infarction, acute coronary syndrome, transient ischemic attack, or stroke within 3 months prior to randomization.
10. Revascularization therapy (coronary artery bypass grafting, percutaneous intervention, or major surgery) within 3 months prior to randomization; or planning cardiac surgery or revascularization.
11. Already receiving erythropoietin, IV or oral iron therapy, and blood transfusion in previous 30 days prior to randomization.
12. Use of concurrent immunosuppressive therapy
13. Any of the following diseases that hinders exercise testing: severe musculoskeletal disease, unstable angina, obstructive cardiomyopathy, severe uncorrected valvular disease, or uncontrolled slow or rapid arrhythmia (mean ventricular rate >100 beats/min at rest), or uncontrolled hypertension with blood pressure >160/100 mm Hg.
14. Investigator considers a possible alternative diagnosis to account for the patient's HF symptoms: severe obesity, primary pulmonary hypertension, or chronic obstructive pulmonary disease.
15. Pregnancy or breast feeding.
16. Participation in another intervention study involving a drug or device within the past 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in peak VO2 (ml/min/kg） | Baseline to Week 52
  Peak VO2 measured by a maximal effort Cardiopulmonary Exercise Test (CPET)

SECONDARY OUTCOMES:
Change in VO2 at ventilatory threshold (ml/min） | Baseline to Week 52
  Measured by CPET
Change in heart rate at peak exercise (bpm) | Baseline to Week 52
  Measured by CPET
Change in peak respiratory exchange ratio | Baseline to Week 52
  Measured by CPET
Change in 6-minute walking distance (m) | Baseline to Week 26 and Week 52
Change in myocardial iron content by cardiac magnetic resonance imaging T2 star | Baseline to Week 52
  Measured by cardiac magnetic resonance imaging
Change in skeletal muscle iron content by magnetic resonance imaging T2 star | Baseline to Week 52
  Measured by skeletal muscle magnetic resonance imaging
Change in the clinical summary score by Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline to Week 52
  The KCCQ is a validated instrument for self-assessment of quality of life and health status in heart failure patients. The clinical summary score, which is derived from the physical limitations and heart failure symptoms domains of the KCCQ is a valid measure for assessing the patient's health aspects that may be influenced by CV medications. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Change in the EQ-5D-5L questionnaire indexed value | Baseline to Week 52
  EQ-5D-5L: European Quality of Life-5 Dimensions-5 Levels The EQ 5D questionnaire consists of a health descriptive system for participants to self-classify and rate their health status on the day of administration. The descriptive system includes 5 items/dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, which are coded from 1 (best state) to 5 (worst state).
Change in cognitive function score by Mini-Mental State Examination (MMSE) | Baseline to Week 52
  The MMSE is a cognitive test. The score is ranged from 0-30 (units of a scale). 30 points is the better outcome. The investigators will assess the change in the score.
Change in concentration of N-terminal pro-brain natriuretic peptide (NT-proBNP, pg/mL) | Baseline to Week 52
  Tested in blood samples
Change in left ventricular ejection fraction (LVEF, %) | Baseline to Week 52
  Assessed by echocardiography
Change in left ventricular global longitudinal stress (LVGLS, %) | Baseline to Week 52
  Assessed by echocardiography
Mortality and heart failure-related hospitalization rates | Up to 52 weeks
  Effects on mortality and HF-related hospitalization rates in patients with heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided